CLINICAL TRIAL: NCT00994890
Title: A MULTICENTRE, RANDOMIZED, DOUBLE-BLIND,LONG TERM STUDY OF THE SAFETY OF SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: A Long Term Study of the Safety of Tanezumab When Administered By Subcutaneous Injections
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A4091043; SC OA SAFETY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Double-blind safety
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — tanezumab; Biological Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tanezumab 2.5 mg (Experimental)
  Interventions: Drug: Tanezumab 2.5 mg
- Tanezumab 5 mg (Experimental)
  Interventions: Drug: Tanezumab 5 mg
- Tanezumab 10 mg (Experimental)
  Interventions: Drug: Tanezumab 10 mg

INTERVENTIONS:
Drug: Tanezumab 2.5 mg — Tanezumab 2.5 mg administered by subcutaneous injection every 8 weeks for a total of 7 injections administered over approximately 1 year
  Other Names: Biological
  Arms: Tanezumab 2.5 mg
Drug: Tanezumab 5 mg — Tanezumab 5 mg administered by subcutaneous injection every 8 weeks for a total of 7 injections administered over approximately 1 year
  Other Names: Biological
  Arms: Tanezumab 5 mg
Drug: Tanezumab 10 mg — Tanezumab 10 mg administered by subcutaneous injection every 8 weeks for a total of 7 injections administered over approximately 1 year
  Other Names: Biological
  Arms: Tanezumab 10 mg

SUMMARY:
This study will investigate the safety of three fixed dose levels of tanezumab (2.5 mg, 5 mg, and 10 mg) administered at an 8-week interval by subcutaneous injection multiple (7) times during the study treatment period.

DETAILED DESCRIPTION:
Safety study of tanezumab in relief of osteoarthritis pain This study was terminated on 6 December 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip based on American College of Rheumatology criteria with a radiographic (X ray) confirmation (a Kellgren Lawrence x-ray grade of ≥2);

Exclusion Criteria:

* Body mass index (BMI) of >39 kg/m2;
* Pregnancy or intent to become pregnant
* Planned surgical procedure during the duration of the study
* History of clinically significant cardiovascular, central nervous system or psychiatric disease
* Previous exposure to exogenous NGF or to an anti NGF antibody;
* Use of biologics other than study medication, Live or live-attenuated intranasal vaccines (eg, Flumist), are allowable exceptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2010-12-07 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (99):
  - Mobile Diagnostic Center, Mobile, Alabama
  - Seton Medical Management, Inc., Mobile, Alabama
  - Phoenix Rheumatology Specialists, Ltd., Phoenix, Arizona
  - Radiant Research, Inc, Scottsdale, Arizona
  - Advanced Arthritis Care and Research, Scottsdale, Arizona
  - Catalina Pointe Clinical Research, Inc, Tucson, Arizona
  - Ft. Smith Rheumatology, PC, Fort Smith, Arkansas
  - Larry Watkins, MD, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - OrthoArkansas, PA, Little Rock, Arkansas
  - Radiology Consultants, Little Rock, Arkansas
  - Medvin Clinical Research, Covina, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - Staywell Research, Northridge, California
  - University Imaging Centers, Northridge, California
  - C Michael Neuwelt, MD, San Leandro, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Medvin Clinical Research, Whittier, California
  - RASF Clinical Research Center, Boca Raton, Florida
  - Sunrise Medical Research, Lauderdale Lake, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - MIMA Century Research Associate, Melbourne, Florida
  - Osler Medical, Inc., Melbourne, Florida
  - Renstar Medical Research, Ocala, Florida
  - American Family Medical, Ocala, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Pensacola Research Consultants, Inc., Pensacola, Florida
  - Radiant Research, Inc, Pinellas Park, Florida
  - Jarred Frydman, DO, Plantation, Florida
  - Orthopaedic Center of South Flordia, Plantation, Florida
  - Advanced Medical Research, Port Orange, Florida
  - Center for Arthritis and Rheumatic Diseases, South Miami, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Radiant Research, Inc, Chicago, Illinois
  - Methodist Medical Group Rheumatology, Peoria, Illinois
  - Methodist Research Administration Office, Peoria, Illinois
  - Rockford Health Physicians, Rockford, Illinois
  - Radiant Research, Inc, Overland Park, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Central Kentucky Research Associates, Mount Sterling, Kentucky
  - Mt. Sterling Clinic, Mount Sterling, Kentucky
  - Boston Clinical Trails, Inc., Boston, Massachusetts
  - Woodrail Clinic, Columbia, Missouri
  - University Physicians, Columbia, Missouri
  - Kansas City Internal Medicine, Lee's Summit, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Advance Clinical Research Inc, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Barbara A. Caciolo, St Louis, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska
  - Radiant Research, Inc, Las Vegas, Nevada
  - Buffalo Rheumatology, Orchard Park, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Robert A. Harrell, MD, Durham, North Carolina
  - Piedmont Imaging, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Radiant Research, Inc, Columbus, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Bone Joint & Spine Surgeons, Inc., Toledo, Ohio
  - McBride Clinic, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Integrated Medical Group PC/Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Research Across America @ Oyster Point Family Health Center, Lancaster, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Allegheny North Arthritis Center, Wexford, Pennsylvania
  - Jeffry A. Lindenbaum D.O., P.C., Yardley, Pennsylvania
  - Anderson Radiology, Anderson, South Carolina
  - Primary Care Associates, Anderson, South Carolina
  - Radiant Research, Inc., Anderson, South Carolina
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute, LLC, Germantown, Tennessee
  - Wolf River Medical Group. LLC, Germantown, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Office of John M. Joseph, M.D., Carrollton, Texas
  - Arthritis Care and Diagnostic Center, Dallas, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Nothwest Diagonstic Clinic, PA, Houston, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
  - Texas Research Center, LP, Sugar Land, Texas
  - Trinity Clinic, Office of Research Administration, Tyler, Texas
  - Trinity Clinic, Rheumatology, Tyler, Texas
  - Physicians' Research Options, LLC, Draper, Utah
  - Lone Peak Family Medicine, Draper, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Arthritis and Rheumatic Disease Associates, PC, Burke, Virginia
  - Alan E. Schulman, MD, Richmond, Virginia
  - Steven Maestrello, M.D., Richmond, Virginia
  - Richard Neiman, MD Inc., Kirkland, Washington
  - South Puget Sound Clinical Research Center, Olympia, Washington
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin
  - Arthritis Clinic, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091043&StudyName=A%20Long%20Term%20Study%20of%20the%20Safety%20of%20Tanezumab%20When%20Administered%20By%20Subcutaneous%20Injections

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to United States Food and Drug Administration (FDA) imposed clinical hold, study was terminated prematurely and a maximum of only 4 doses of the 7 planned doses of tanezumab (RN624 or PF-04383119) subcutaneous injection were administered in the study.
Groups:
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 milligram (mg) injection subcutaneously every 8 weeks up to 24 weeks.
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection subcutaneously every 8 weeks up to 24 weeks.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg injection subcutaneously every 8 weeks up to 24 weeks.
Period: Overall Study
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Started | 231 | 222 | 226
Treated | 230 | 222 | 226
Completed | 0 | 0 | 0
Not Completed | 231 | 222 | 226
Not completed — Adverse Event | 13 | 9 | 11
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 6 | 1 | 3
Not completed — No longer willing to participate | 8 | 5 | 13
Not completed — Protocol Violation | 2 | 4 | 0
Not completed — Study terminated by sponsor | 199 | 201 | 197
Not completed — Randomized, but not treated | 1 | 0 | 0
Not completed — Other | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg | Total
Number analyzed (Participants) | 230 | 222 | 226 | 678
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 11 | 7 | 4 | 22
  45 to 64 years | 128 | 124 | 113 | 365
  Greater than or equal to (>=) 65 years | 91 | 91 | 109 | 291
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 157 | 161 | 470
  Male | 78 | 65 | 65 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 112 days after last dose of study medication (up to 345 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants
  AEs | 158 | 169 | 181
  SAEs | 17 | 12 | 20

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory analysis included blood chemistry, hematology, urinalysis and pregnancy test.
Time Frame: Baseline to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 221 | 220 | 220
Participants | 136 | 121 | 130

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: All standard intervals (PR, QRS, QT, QT interval corrected for heart rate using Fridericia's formula [QTcF], QT interval corrected for heart rate using Bazett's formula [QTcB], RR intervals and heart rate) were analyzed. Participants with abnormal ECG findings reported as adverse events were presented.
Time Frame: Baseline up to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants
  Atrioventricular block first degree | 0 | 1 | 0
  Bundle branch block right | 0 | 0 | 1
  Supraventricular extrasystoles | 0 | 0 | 1
  Supraventricular tachycardia | 0 | 1 | 0
  Tachycardia | 1 | 1 | 2
  ECG QRS complex prolonged | 1 | 0 | 0
  ECG T wave abnormal | 0 | 1 | 0
  ECG T wave inversion | 1 | 0 | 1

4. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 2
Description: NIS: 74-item, assess cranial nerves, muscle weakness, reflexes, sensation; scored separately for left, right limbs (37 items for each). Cranial nerves included 5 items (3rd nerve, 6th nerve, facial weakness, palate weakness, tongue weakness), muscle weakness included 19 items (respiratory,neck flexion, shoulder abduction, elbow flexion, brachioradialis,elbow extension, wrist flexion,wrist extension,finger flexion,finger spread,thumb abduction,hip flexion,hip extension,knee flexion,knee extension,ankle dorsiflexors,ankle plantar flexors,toe extensors,toe flexors), each item scored on scale 0=normal to 4=paralysis, higher score=greater weakness. Reflexes included 5 items (quadriceps femoris, triceps surae, biceps brachii, triceps brachii, brachioradialis), sensation included 4 items each for great toe and index finger (touch pressure, pin prick, vibration, joint position), each item scored as 0=normal, 1=decreased, 2=absent. Total NIS score range 0-244, higher score=greater impairment.
Time Frame: Baseline, Week 2
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 229 | 222 | 225
units on a scale
  Baseline | 2.04 (3.93) | 1.52 (3.17) | 1.76 (3.53)
  Change at Week 2: number analyzed (Participants) | 223 | 218 | 218
  Change at Week 2 | -0.43 (1.51) | -0.36 (2.04) | -0.23 (1.78)

5. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 4
Description: as for outcome 4
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 218 | 215 | 218
units on a scale | -0.35 (1.72) | -0.15 (2.12) | -0.10 (1.83)

6. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 8
Description: as for outcome 4
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 215 | 216 | 216
units on a scale | -0.39 (2.10) | -0.08 (2.30) | -0.34 (2.14)

7. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 16
Description: as for outcome 4
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 188 | 207 | 203
units on a scale | -0.60 (2.24) | -0.17 (2.66) | -0.24 (2.61)

8. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 161 | 176 | 165
units on a scale | -0.46 (2.14) | -0.38 (2.53) | -0.19 (2.44)

9. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 32
Description: as for outcome 4
Time Frame: Baseline, Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 81 | 90 | 91
units on a scale | -0.72 (2.15) | -0.11 (2.26) | -0.34 (3.02)

10. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 40
Description: as for outcome 4
Time Frame: Baseline, Week 40
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 22 | 23 | 27
units on a scale | -0.82 (2.11) | -0.39 (1.41) | 0.00 (3.98)

11. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 48
Description: as for outcome 4
Time Frame: Baseline, Week 48
Population: ITT analysis set. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. Results are not reported for Tanezumab 5 mg group because all participants in this group had discontinued the study before Week 48.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 1 | 0 | 1
units on a scale | -2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable in this group. |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable in this group.

12. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Findings
Description: Physical examination included examination of abdomen, ears, extremities, eyes, head, heart, lungs, lymph nodes, neck, nose, skin, throat, thyroid, muscoskeletal, neurological and peripheral vascular system.
Time Frame: Baseline to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants | 13 | 13 | 18

13. Primary Outcome: Number of Participants With Anti-Drug Antibody (ADA) at Day 1
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure at any time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 215 | 213 | 208
Participants | 1 | 1 | 1

14. Primary Outcome: Number of Participants With Anti-Drug Antibody (ADA) at Week 8
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative ELISA.
Time Frame: Week 8
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 206 | 204 | 203
Participants | 1 | 2 | 1

15. Primary Outcome: Number of Participants With Anti-Drug Antibody (ADA) at Week 24
Description: as for outcome 14
Time Frame: Week 24
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 78 | 93 | 82
Participants | 0 | 1 | 0

16. Primary Outcome: Number of Participants With Anti-Drug Antibody (ADA) at Week 50
Description: as for outcome 14
Time Frame: Week 50
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 171 | 176 | 172
Participants | 3 | 3 | 1

17. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Examination of vital signs included body temperature, systolic blood pressure, diastolic blood pressure, pulse rate and respiratory rate. Participants with abnormal vital sign findings reported as adverse events were presented.
Time Frame: Baseline up to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants
  Blood pressure increased | 0 | 3 | 1
  Hypertension | 8 | 4 | 5
  Hypotension | 0 | 0 | 1

18. Primary Outcome: Number of Participants With Injection-Site Reactions at Day 1
Description: Assessment of the injection-site reactions were based on presence of erythema (redness), induration (swelling), ecchymosis (bruising), pruritus (itching) and pain that occurred after the injection had been administered (not related to pain of needle insertion).
Time Frame: Day 1
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants | 9 | 12 | 9

19. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 2
Description: as for outcome 18
Time Frame: Week 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 221 | 218 | 219
Participants | 7 | 3 | 4

20. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 4
Description: as for outcome 18
Time Frame: Week 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 219 | 212 | 218
Participants | 1 | 1 | 1

21. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 8
Description: as for outcome 18
Time Frame: Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 186 | 191 | 192
Participants | 4 | 6 | 7

22. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 16
Description: as for outcome 18
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 107 | 123 | 113
Participants | 2 | 1 | 1

23. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 24
Description: as for outcome 18
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 54 | 67 | 64
Participants | 1 | 0 | 0

24. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 32
Description: as for outcome 18
Time Frame: Week 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 31 | 28 | 32
Participants | 0 | 0 | 0

25. Primary Outcome: Number of Participants With Injection-Site Reactions at Week 40
Description: as for outcome 18
Time Frame: Week 40
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 11 | 11 | 12
Participants | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or index hip during past 48 hours. It was calculated as mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 to 10, where higher scores indicated higher pain.
Time Frame: Baseline, Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: ITT analysis set. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. Missing data was imputed using last observation carried forward (LOCF) method. Due to implementation of the FDA clinical hold, all ongoing participants were discontinued from treatment and did not have an opportunity to complete the 56-week treatment period and no efficacy data beyond the Week 32 visit (i.e., Weeks 40, 48 and 56) was collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 222
units on a scale
  Baseline | 6.35 (1.48) | 6.48 (1.56) | 6.30 (1.48)
  Change at Week 2 | -2.01 (2.02) | -1.97 (2.18) | -1.61 (2.00)
  Change at Week 4 | -2.43 (2.11) | -2.68 (2.15) | -2.50 (2.02)
  Change at Week 8 | -2.20 (2.14) | -2.76 (2.25) | -2.71 (2.14)
  Change at Week 16 | -2.18 (2.25) | -2.85 (2.32) | -2.71 (2.15)
  Change at Week 24 | -2.16 (2.29) | -2.84 (2.31) | -2.69 (2.17)
  Change at Week 32 | -2.15 (2.26) | -2.82 (2.32) | -2.66 (2.14)

27. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint and index hip during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on NRS of 0 to 10, with higher scores indicated worse function. Total score range for WOMAC physical function subscale score was 0 to 10, where higher scores indicated worse function.
Time Frame: Baseline, Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 223
units on a scale
  Baseline | 6.49 (1.54) | 6.58 (1.55) | 6.47 (1.53)
  Change at Week 2 | -2.10 (2.01) | -2.13 (2.15) | -1.92 (1.96)
  Change at Week 4 | -2.50 (2.16) | -2.70 (2.22) | -2.64 (2.09)
  Change at Week 8 | -2.29 (2.10) | -2.83 (2.26) | -2.80 (2.23)
  Change at Week 16 | -2.28 (2.20) | -2.89 (2.35) | -2.84 (2.22)
  Change at Week 24 | -2.26 (2.23) | -2.89 (2.37) | -2.84 (2.21)
  Change at Week 32 | -2.23 (2.22) | -2.90 (2.36) | -2.79 (2.20)

28. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 2, 4, 8,16, 24, 32, 40, 48 and 56
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee (or hip) affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good (no symptom and limitation of normal activities) and 5 = very poor (very severe symptoms and inability to carry out normal activities).
Time Frame: Baseline, Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 228 | 222 | 225
units on a scale
  Baseline | 3.38 (0.59) | 3.36 (0.57) | 3.32 (0.53)
  Change at Week 2 | -0.70 (0.78) | -0.64 (0.85) | -0.64 (0.84)
  Change at Week 4 | -0.85 (0.79) | -0.86 (0.86) | -0.77 (0.87)
  Change at Week 8 | -0.72 (0.80) | -0.83 (0.83) | -0.82 (0.92)
  Change at Week 16 | -0.69 (0.83) | -0.84 (0.86) | -0.80 (0.91)
  Change at Week 24 | -0.71 (0.87) | -0.82 (0.88) | -0.80 (0.88)
  Change at Week 32 | -0.69 (0.88) | -0.82 (0.88) | -0.80 (0.88)

29. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: OMERACT-OARSI response: greater than or equal to (>=) 50 percent (%) improvement from baseline and absolute change from baseline of >=2 units in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 223
percentage of participants
  Week 2 | 57.8 [51 to 64] | 58.6 [52 to 65] | 49.3 [43 to 56]
  Week 4 | 64.9 [59 to 71] | 70.5 [64 to 76] | 73.5 [68 to 79]
  Week 8 | 61.8 [55 to 68] | 68.6 [63 to 75] | 70.9 [65 to 77]
  Week 16 | 59.1 [53 to 66] | 68.6 [63 to 75] | 72.2 [66 to 78]
  Week 24 | 58.7 [52 to 65] | 68.2 [62 to 74] | 71.7 [66 to 78]
  Week 32 | 58.2 [52 to 65] | 68.2 [62 to 74] | 71.7 [66 to 78]

30. Secondary Outcome: Percentage of Participants With At Least 30 Percent (%), 50%, 70% and 90% Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: Percentage of participants with at least 30%, 50%, 70% and 90% reduction from baseline in WOMAC pain subscale score are reported. WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or index hip during past 48 hours. It was calculated as mean of the scores from the 5 individual questions scored on a 0 to 10 NRS, where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicated higher pain.
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 222
percentage of participants
  Week 2: at least 30% reduction | 48.9 [42 to 55] | 49.1 [42 to 56] | 41.4 [35 to 48]
  Week 2: at least 50% reduction | 28.4 [23 to 34] | 31.4 [25 to 37] | 23.9 [18 to 29]
  Week 2: at least 70% reduction | 13.8 [9 to 18] | 16.8 [12 to 22] | 14.0 [9 to 19]
  Week 2: at least 90% reduction | 4.9 [2 to 8] | 3.6 [1 to 6] | 3.6 [1 to 6]
  Week 4: at least 30% reduction | 57.3 [51 to 64] | 62.7 [56 to 69] | 60.4 [54 to 67]
  Week 4: at least 50% reduction | 39.1 [33 to 45] | 40.9 [34 to 47] | 41.0 [35 to 47]
  Week 4: at least 70% reduction | 21.3 [16 to 27] | 24.5 [19 to 30] | 22.5 [17 to 28]
  Week 4: at least 90% reduction | 7.6 [4 to 11] | 6.8 [3 to 10] | 6.3 [3 to 10]
  Week 8: at least 30% reduction | 50.7 [44 to 57] | 62.7 [56 to 69] | 66.2 [60 to 72]
  Week 8: at least 50% reduction | 35.1 [29 to 41] | 46.4 [40 to 53] | 46.4 [40 to 53]
  Week 8: at least 70% reduction | 18.2 [13 to 23] | 26.8 [21 to 33] | 27.0 [21 to 33]
  Week 8: at least 90% reduction | 7.6 [4 to 11] | 11.4 [7 to 16] | 10.8 [7 to 15]
  Week 16: at least 30% reduction | 52.4 [46 to 59] | 62.3 [56 to 69] | 65.3 [59 to 72]
  Week 16: at least 50% reduction | 37.3 [31 to 44] | 50.0 [43 to 57] | 45.5 [39 to 52]
  Week 16: at least 70% reduction | 20.4 [15 to 26] | 28.6 [23 to 35] | 28.4 [22 to 34]
  Week 16: at least 90% reduction | 6.2 [3 to 9] | 11.8 [8 to 16] | 12.2 [8 to 16]
  Week 24: at least 30% reduction | 50.2 [44 to 57] | 62.7 [56 to 69] | 65.3 [59 to 72]
  Week 24: at least 50% reduction | 37.3 [31 to 44] | 50.0 [43 to 57] | 45.5 [39 to 52]
  Week 24: at least 70% reduction | 20.4 [15 to 26] | 28.2 [22 to 34] | 28.8 [23 to 35]
  Week 24: at least 90% reduction | 7.1 [4 to 10] | 11.8 [8 to 16] | 11.7 [7 to 16]
  Week 32: at least 30% reduction | 51.1 [45 to 58] | 62.3 [56 to 69] | 64.9 [59 to 71]
  Week 32: at least 50% reduction | 36.9 [31 to 43] | 49.5 [43 to 56] | 44.1 [38 to 51]
  Week 32: at least 70% reduction | 20.4 [15 to 26] | 27.7 [22 to 34] | 27.9 [22 to 34]
  Week 32: at least 90% reduction | 6.7 [3 to 10] | 11.4 [7 to 16] | 11.3 [7 to 15]

31. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index knee or index hip during past 48 hours. It is calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline at Week 16 are reported.
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 115 | 135 | 118
percentage of participants
  Week 16: greater than (>) 0% | 82.6 | 85.2 | 89.0
  Week 16: >=10% | 74.8 | 81.5 | 82.2
  Week 16: >=20% | 65.2 | 71.9 | 73.7
  Week 16: >=30% | 58.3 | 63.0 | 67.8
  Week 16: >=40% | 47.0 | 57.0 | 60.2
  Week 16: >=50% | 43.5 | 51.9 | 50.0
  Week 16: >=60% | 33.0 | 41.5 | 41.5
  Week 16: >=70% | 28.7 | 32.6 | 33.9
  Week 16: >=80% | 18.3 | 21.5 | 22.9
  Week 16: >=90% | 9.6 | 14.8 | 14.4
  Week 16: 100% | 4.3 | 3.7 | 5.9

32. Secondary Outcome: Percentage of Participants With Improvement of At Least 2 Points in Patient Global Assessment (PGA) of Osteoarthritis
Description: Participants answered: "Considering all the ways your osteoarthritis in your knee (or hip) affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good and 5 = very poor. Improvement signifies a decrease of at least 2 points on the 5-point scale relative to baseline value.
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 228 | 222 | 225
percentage of participants
  Week 2 | 14.5 [10 to 19] | 15.8 [11 to 21] | 13.3 [9 to 18]
  Week 4 | 20.2 [15 to 25] | 20.3 [15 to 26] | 16.9 [12 to 22]
  Week 8 | 15.8 [11 to 21] | 18.9 [14 to 24] | 24.9 [19 to 31]
  Week 16 | 15.4 [11 to 20] | 18.0 [13 to 23] | 20.9 [16 to 26]
  Week 24 | 16.7 [12 to 22] | 18.5 [13 to 24] | 20.0 [15 to 25]
  Week 32 | 16.2 [11 to 21] | 18.5 [13 to 24] | 20.0 [15 to 25]

33. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in index knee or index hip during past 48 hours. It is calculated as mean of the scores from 2 individual questions scored on NRS of 0 to 10, with higher scores indicate higher stiffness. Total score range for WOMAC stiffness subscale score is 0 to 10, where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of knee or hip.
Time Frame: Baseline, Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 223
units on a scale
  Baseline | 6.78 [6.55 to 7.01] | 6.85 [6.61 to 7.08] | 6.73 [6.50 to 6.95]
  Change at Week 2 | -2.32 [-2.63 to -2.02] | -2.42 [-2.75 to -2.10] | -2.29 [-2.61 to -1.98]
  Change at Week 4 | -2.73 [-3.05 to -2.40] | -3.01 [-3.34 to -2.68] | -2.99 [-3.31 to -2.67]
  Change at Week 8 | -2.43 [-2.75 to -2.10] | -3.17 [-3.50 to -2.84] | -3.05 [-3.41 to -2.69]
  Change at Week 16 | -2.43 [-2.76 to -2.10] | -3.20 [-3.54 to -2.87] | -3.15 [-3.50 to -2.80]
  Change at Week 24 | -2.41 [-2.75 to -2.07] | -3.20 [-3.54 to -2.86] | -3.10 [-3.45 to -2.75]
  Change at Week 32 | -2.36 [-2.70 to -2.03] | -3.21 [-3.55 to -2.87] | -3.05 [-3.40 to -2.71]

34. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee or hip. Each item was scored on a 0 to 10 NRS scale, where higher scores indicated higher pain/stiffness or worse function. WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranged from 0 to 10, where higher score indicated worse response.
Time Frame: Baseline, Week 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 223
units on a scale
  Baseline | 6.54 (1.45) | 6.64 (1.50) | 6.50 (1.41)
  Change at Week 2 | -2.14 (1.99) | -2.18 (2.13) | -1.94 (1.96)
  Change at Week 4 | -2.56 (2.14) | -2.80 (2.18) | -2.71 (2.05)
  Change at Week 8 | -2.31 (2.11) | -2.92 (2.24) | -2.85 (2.23)
  Change at Week 16 | -2.30 (2.21) | -2.98 (2.29) | -2.90 (2.22)
  Change at Week 24 | -2.27 (2.26) | -2.97 (2.32) | -2.88 (2.21)
  Change at Week 32 | -2.25 (2.23) | -2.98 (2.31) | -2.83 (2.20)

35. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item: Pain When Walking on a Flat Surface at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: Participants answered: "How much pain have you had when walking on a flat surface?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 220 | 222
units on a scale
  Baseline | 6.15 (1.86) | 6.32 (1.84) | 6.20 (1.86)
  Change at Week 2 | -1.95 (2.17) | -1.94 (2.38) | -1.67 (2.34)
  Change at Week 4 | -2.26 (2.31) | -2.59 (2.34) | -2.45 (2.29)
  Change at Week 8 | -2.03 (2.42) | -2.65 (2.50) | -2.63 (2.32)
  Change at Week 16 | -2.00 (2.54) | -2.66 (2.48) | -2.57 (2.46)
  Change at Week 24 | -1.96 (2.55) | -2.65 (2.51) | -2.60 (2.42)
  Change at Week 32 | -1.96 (2.51) | -2.63 (2.51) | -2.56 (2.43)

36. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item: Pain When Going Up or Down Stairs at Week 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: Participants answered: "How much pain have you had when going up or down the stairs?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 224 | 219 | 222
units on a scale
  Baseline | 7.52 (1.64) | 7.64 (1.68) | 7.54 (1.72)
  Change at Week 2 | -2.34 (2.28) | -2.25 (2.43) | -1.99 (2.30)
  Change at Week 4 | -2.86 (2.58) | -3.01 (2.47) | -2.77 (2.45)
  Change at Week 8 | -2.60 (2.48) | -3.03 (2.59) | -3.01 (2.53)
  Change at Week 16 | -2.51 (2.63) | -3.05 (2.67) | -3.01 (2.62)
  Change at Week 24 | -2.47 (2.66) | -3.00 (2.67) | -2.98 (2.55)
  Change at Week 32 | -2.46 (2.63) | -3.01 (2.66) | -2.94 (2.54)

37. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
days | NA [NA to NA] — Median and full range were not evaluable since no participant discontinued due to lack of efficacy. | NA [NA to NA] — Median and full range were not evaluable since no participant discontinued due to lack of efficacy. | NA [82.0 to 82.0] — Median was not evaluable since only 1 participant discontinued due to lack of efficacy.

38. Secondary Outcome: Number of Participants Who Discontinued Due to Lack of Efficacy
Time Frame: Baseline up to Week 50
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants | 0 | 0 | 1

39. Secondary Outcome: Percentage of Participants Who Used Concomitant Analgesic Medication
Description: United States Food and Drug Administration (FDA) approved analgesics were permitted as concomitant medications to relieve the pain of osteoarthritis. These medications included opioids, topical analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), capsaicin products and viscosupplementation (example, hyaluronan) and were prescribed at the discretion of the Investigator.
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: ITT analysis set. 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group. Data were not collected beyond Week 48 due to premature termination of the study in response to FDA clinical hold.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 219 | 221
percentage of participants
  Week 2: number analyzed (Participants) | 225 | 219 | 219
  Week 2 | 53.8 [47 to 60] | 49.8 [43 to 56] | 52.5 [46 to 59]
  Week 4: number analyzed (Participants) | 223 | 216 | 221
  Week 4 | 52.9 [46 to 59] | 47.7 [41 to 54] | 51.6 [45 to 58]
  Week 8: number analyzed (Participants) | 216 | 217 | 221
  Week 8 | 53.7 [47 to 60] | 47.9 [41 to 55] | 51.6 [45 to 58]
  Week 16: number analyzed (Participants) | 162 | 178 | 182
  Week 16 | 50.6 [43 to 58] | 47.8 [40 to 55] | 50.5 [43 to 58]
  Week 24: number analyzed (Participants) | 93 | 98 | 88
  Week 24 | 49.5 [39 to 60] | 49.0 [39 to 59] | 48.9 [38 to 59]
  Week 32: number analyzed (Participants) | 18 | 21 | 23
  Week 32 | 33.3 [12 to 55] | 47.6 [26 to 69] | 52.2 [32 to 73]
  Week 40: number analyzed (Participants) | 1 | 1 | 1
  Week 40 | 100 [100 to 100] | 0 [0 to 0] | 100 [100 to 100]
  Week 48: number analyzed (Participants) | 0 | 1 | 0
  Week 48 |  | 0 [0 to 0] |

40. Secondary Outcome: Days Per Week of Concomitant Analgesic Medication Usage
Description: United States FDA-approved analgesics were permitted as concomitant medications to relieve the pain of OA. These medications included opioids, topical analgesics, NSAIDs, capsaicin products and viscosupplementation (example, hyaluronan) and were prescribed at the discretion of the Investigator.
Time Frame: Week 2, 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: ITT analysis set. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group. Data were not collected beyond Week 48 due to premature termination of the study in response to FDA clinical hold.
Measure: Median (Full Range); unit: days per week
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 225 | 219 | 221
days per week
  Week 2: number analyzed (Participants) | 225 | 219 | 219
  Week 2 | 7.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 7.0 [0.0 to 7.0]
  Week 4: number analyzed (Participants) | 223 | 216 | 221
  Week 4 | 7.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 7.0 [0.0 to 7.0]
  Week 8: number analyzed (Participants) | 216 | 217 | 221
  Week 8 | 7.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 2.9 [0.0 to 7.0]
  Week 16: number analyzed (Participants) | 162 | 178 | 182
  Week 16 | 2.5 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.4 [0.0 to 7.0]
  Week 24: number analyzed (Participants) | 93 | 98 | 88
  Week 24 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0]
  Week 32: number analyzed (Participants) | 18 | 21 | 23
  Week 32 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 7.0 [0.0 to 7.0]
  Week 40: number analyzed (Participants) | 1 | 1 | 1
  Week 40 | 7.0 [7.0 to 7.0] | 0.0 [0.0 to 0.0] | 7.0 [7.0 to 7.0]
  Week 48: number analyzed (Participants) | 0 | 1 | 0
  Week 48 |  | 0.0 [0.0 to 0.0] |

41. Other Pre Specified Outcome: Number of Participants With Subcutaneous Doses of Study Medication
Description: Number of participants are reported based on the maximum number of subcutaneous doses of study medication received.
Time Frame: Day 1 up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of subcutaneous study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Number analyzed (Participants) | 230 | 222 | 226
Participants
  1 dose | 48 | 36 | 38
  2 doses | 99 | 89 | 103
  3 doses | 64 | 72 | 61
  4 doses | 19 | 25 | 24

ADVERSE EVENTS:
Description: Cases of osteonecrosis (ON) reported in this and other A409 studies conducted up to 2010 were adjudicated post-hoc by an expert committee(2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492
Arm/Group | Tanezumab 2.5 mg | Tanezumab 5 mg | Tanezumab 10 mg
Serious Adverse Events (participants affected / at risk) | 17/230 | 12/222 | 20/226
Other Adverse Events (participants affected / at risk) | 132/230 | 137/222 | 153/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=230) | Tanezumab 5 mg (N=222) | Tanezumab 10 mg (N=226)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 2.5 mg (N=230) | Tanezumab 5 mg (N=222) | Tanezumab 10 mg (N=226)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6
Nausea (Gastrointestinal disorders) | 6 | 6 | 11
Fatigue (General disorders) | 3 | 0 | 8
Injection site reaction (General disorders) | 19 | 21 | 20
Oedema peripheral (General disorders) | 9 | 16 | 22
Bronchitis (Infections and infestations) | 6 | 9 | 7
Nasopharyngitis (Infections and infestations) | 3 | 5 | 6
Sinusitis (Infections and infestations) | 6 | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 12 | 9 | 12
Urinary tract infection (Infections and infestations) | 11 | 12 | 20
Contusion (Injury, poisoning and procedural complications) | 4 | 1 | 5
Fall (Injury, poisoning and procedural complications) | 7 | 5 | 12
Joint injury (Injury, poisoning and procedural complications) | 3 | 6 | 6
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 5
Blood creatine phosphokinase increased (Investigations) | 6 | 8 | 9
Blood lactate dehydrogenase increased (Investigations) | 1 | 5 | 3
Blood triglycerides increased (Investigations) | 1 | 5 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 30 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 | 10 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 15 | 12
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 11 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 12 | 16
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 1 | 9
Burning sensation (Nervous system disorders) | 1 | 5 | 2
Carpal tunnel syndrome (Nervous system disorders) | 8 | 3 | 7
Dizziness (Nervous system disorders) | 3 | 5 | 8
Headache (Nervous system disorders) | 9 | 6 | 10
Hypoaesthesia (Nervous system disorders) | 14 | 6 | 15
Paraesthesia (Nervous system disorders) | 13 | 17 | 25
Anxiety (Psychiatric disorders) | 5 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 6 | 1
Hypertension (Vascular disorders) | 8 | 4 | 5

LIMITATIONS AND CAVEATS:
Due to United States FDA imposed clinical hold, enrollment was stopped and study was terminated prematurely. Due to this, injection-site reaction data were not collected beyond Week 40 and NIS data were not collected beyond Week 48.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.